CLINICAL TRIAL: NCT02891408
Title: A Phase 1 Open-Label, Parallel-Group, Single-Dose Study to Evaluate the Pharmacokinetics of GS-0976 or Fenofibrate in Subjects With Normal and Impaired Hepatic Function
Brief Title: Study to Evaluate the Pharmacokinetics of Firsocostat or Fenofibrate in Adults With Normal and Impaired Hepatic Function
Acronym: HI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-426-3988
Record Dates: First submitted 2016-09-01; First posted 2016-09-07 (Estimated); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Nonalcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — firsocostat; Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg (Experimental): Participants with mild hepatic impairment will receive a single dose of firsocostat 20 mg (2 × 10 mg capsules).
  Interventions: Drug: Firsocostat
- Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg (Experimental): Matched normal hepatic function participants to mild hepatic impairment participants will receive a single dose of firsocostat 20 mg (2 × 10 mg capsules).
  Interventions: Drug: Firsocostat
- Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg (Experimental): Participants with moderate hepatic impairment will receive a single dose of firsocostat 20 mg (2 × 10 mg capsules).
  Interventions: Drug: Firsocostat
- Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg (Experimental): Matched normal hepatic function participants to moderate hepatic impairment participants will receive a single dose of firsocostat 20 mg (2 × 10 mg capsules).
  Interventions: Drug: Firsocostat
- Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg (Experimental): Participants with severe hepatic impairment will receive a single dose of firsocostat 5 mg (1 × 5 mg capsule).
  Interventions: Drug: Firsocostat
- Cohort 3 (Normal Hepatic Function) Firsocostat 5 mg (Experimental): Matched normal hepatic function participants to severe hepatic impairment participants will receive a single dose of firsocostat 5 mg (1 × 5 mg capsule).
  Interventions: Drug: Firsocostat
- Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg (Experimental): Participants with mild hepatic impairment will receive a single dose of fenofibrate 48 mg (1 × 48 mg tablet).
  Interventions: Drug: Fenofibrate
- Cohort 4 (Normal Hepatic Function) Fenofibrate 48 mg (Experimental): Matched normal hepatic function participants to mild hepatic impairment participants, will receive a single dose of fenofibrate 48 mg (1 × 48 mg tablet).
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: Firsocostat — Capsule(s) administered orally on Day 1
  Other Names: GS-0976
  Arms: Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg; Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg; Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg; Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg; Cohort 3 (Normal Hepatic Function) Firsocostat 5 mg; Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg
Drug: Fenofibrate — Tablet administered orally on Day 1
  Arms: Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg; Cohort 4 (Normal Hepatic Function) Fenofibrate 48 mg

SUMMARY:
The primary objectives of this study are to evaluate the single-dose pharmacokinetics (PK) of firsocostat in adults with normal hepatic function, and mild, moderate, or severe hepatic impairment and to evaluate the single-dose PK of fenofibrate in adults with normal hepatic function and mild hepatic impairment.

ELIGIBILITY:
Key Inclusion Criteria:

Cohort 1 (Mild Hepatic Impairment):

* Male and non-pregnant/non-lactating females with mildly impaired and normal hepatic function.
* Individuals will be current non-smokers (no use of tobacco, nicotine-containing or tetrahydrocannabinol (THC)-containing products within the last 14 days).
* Each individual in the control group will be matched for age (± 10 years), gender, race, and body mass index (± 15% 18 ≤ body mass index (BMI) ≤ 36 kg/m^2) with an individual in the mild hepatic impairment group.
* Individuals with mild hepatic impairment must have a score of 5-6 on the Child-Pugh-Turcotte (CPT) Classification at screening, have diagnosis of chronic (> 6 months), and stable hepatic impairment with no clinically significant changes within 3 months (or 90 days) prior to study drug administration (Day 1).

Cohort 2 (Moderate Hepatic Impairment):

* Male and non-pregnant/non-lactating females with moderately impaired and normal hepatic function.
* Individuals will be current non-smokers (no smoking of tobacco, nicotine-containing or THC-containing products within the last 14 days).
* Each individual in the control group will be matched for age (± 10 years), gender, race, and body mass index (± 15% 18 ≤ BMI ≤ 36 kg/m^2) with an individual in the moderate hepatic impairment group.
* Individuals with moderate hepatic impairment must have a score of 7-9 on the CPT Classification at screening, have diagnosis of chronic (> 6 months), and stable hepatic impairment with no clinically significant changes within 3 months (or 90 days) prior to study drug administration (Day 1).

Cohort 3 (Severe Hepatic Impairment):

* Male and nonpregnant/non-lactating females with severely impaired and normal hepatic function.
* Individuals will be current non-smokers (no use of tobacco, nicotine-containing or THC-containing products within the last 14 days).
* Each individual in the control group will be matched for age (± 10 years), gender, race, and body mass index (± 15% 18 ≤ BMI ≤ 36 kg/m^2) with an individual in the severe hepatic impairment group.
* Individuals with severe hepatic impairment must have a score of 10-15 on the CPT Classification at screening, have diagnosis of chronic (> 6 months), and stable hepatic impairment with no clinically significant changes within 3 months (or 90 days) prior to study drug administration (Day 1).

Cohort 4 (Mild Hepatic Impairment):

* Male and non-pregnant/non-lactating females with mildly impaired and normal hepatic function.
* Individuals will be current non-smokers (no use of tobacco, nicotine-containing or THC-containing products within the last 14 days).
* Each individual in the control group will be matched for age (± 10 years), gender, race, and body mass index (± 15% 18 ≤ body mass index (BMI) ≤ 36 kg/m^2) with an individual in the mild hepatic impairment group.
* Individuals with mild hepatic impairment must have a score of 5-6 on the Child-Pugh-Turcotte (CPT) Classification at screening, have diagnosis of chronic (> 6 months), and stable hepatic impairment with no clinically significant changes within 3 months (or 90 days) prior to study drug administration (Day 1).

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2016-09-23 (Actual); Primary Completion 2019-05-05 (Actual); Study Completion 2019-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (5):
- United States (5):
  - Tustin, California
  - Miami, Florida
  - Orlando, Florida
  - Minneapolis, Minnesota
  - San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nelson C, Weber E, Yue MS, Millward V, Qin AR, Marbury TC, et al. The Pharmacokinetics of GS-0976, an Acetyl-CoA Carboxylase (ACC) Inhibitor, in Subjects with Mild, Moderate, and Severe Hepatic Impairment [Abstract 1719]. Hepatology AASLD Abstracts 2018;68 (Suppl 1):979A-80A.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in United States. The first participant was screened on 23 September 2016. The last study visit occurred on 13 May 2019.
Pre-assignment Details: In the control groups (normal hepatic function), each participant was matched for age, gender, race, and body mass index with a participant in the hepatic impairment group. 14 total unique participants with normal hepatic function were enrolled in Cohort 1 (N = 10) and Cohort 2 (N = 4). 6 participants with normal hepatic function from Cohort 1 also served as matched controls in Cohort 2.
Groups:
- Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg: Participants with mild hepatic impairment received a single dose of firsocostat 20 mg (2 × 10 mg capsules) orally on Day 1.
- Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg: Participants with moderate hepatic impairment received a single dose of firsocostat 20 mg (2 × 10 mg capsules) orally on Day 1.
- Cohort 1 & 2 (Normal Hepatic Function): Firsocostat 20 mg: Matched normal hepatic function participants to mild or moderate hepatic impairment participants received a single dose of firsocostat 20 mg (2 × 10 mg capsules) orally on Day 1
- Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg: Participants with severe hepatic impairment received a single dose of firsocostat 5 mg (1 × 5 mg capsule) orally on Day 1.
- Cohort 3 (Normal Hepatic Function) Firsocostat 5 mg: Matched normal hepatic function participants to severe hepatic impairment participants received a single dose of firsocostat 5 mg (1 × 5 mg capsule) orally on Day 1.
- Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg: Participants with mild hepatic impairment received a single dose of fenofibrate 48 mg (1 × 48 mg tablet) orally on Day 1.
- Cohort 4 (Normal Hepatic Function) Fenofibrate 48 mg: Matched normal hepatic function participants to mild hepatic impairment participants, received a single dose of fenofibrate 48 mg (1 × 48 mg tablet) orally on Day 1.
Period: Overall Study
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 1 & 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function) Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function) Fenofibrate 48 mg
Started | 10 | 10 | 14 | 10 | 10 | 10 | 10
Completed | 10 | 10 | 13 | 10 | 10 | 10 | 10
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 1 & 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function) Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function) Fenofibrate 48 mg | Total
Number analyzed (Participants) | 10 | 10 | 14 | 10 | 10 | 10 | 10 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (8.1) | 56 (9.1) | 55 (8.0) | 53 (10.8) | 54 (8.4) | 58 (6.4) | 58 (5.1) | 55 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 3 | 4 | 4 | 3 | 3 | 22
  Male | 8 | 7 | 11 | 6 | 6 | 7 | 7 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 7 | 6 | 6 | 6 | 6 | 40
  Not Hispanic or Latino | 7 | 4 | 7 | 4 | 4 | 4 | 4 | 34
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 0 | 4 | 1 | 1 | 2 | 2 | 14
  White | 5 | 9 | 9 | 9 | 9 | 8 | 8 | 57
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUClast of Firsocostat, GS-834773 (Primary Metabolite of Firsocostat), and Fenofibric Acid (Primary Metabolite of Fenofibrate)
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration. The PK of fenofibric acid was evaluated in participants with mild hepatic impairment and matched participants with normal hepatic function (Cohort 4).
Time Frame: Day 1: 0 (predose, ≤ 5 minutes prior to dosing), 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 48, 72, and 96 hours postdose; or 72 hours of early termination from the study (if applicable)
Population: PK Analysis Sets included all enrolled participants who took at least 1 dose of study drug and had at least 1 nonmissing postdose concentration value reported by PK laboratory for corresponding analytes. 6 participants with normal hepatic function served as matched controls across both Cohort 1 and 2.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg: Matched normal hepatic function participants to mild hepatic impairment participants, received a single dose of firsocostat 20 mg (2 × 10 mg capsules) orally on Day 1.
- Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg: Matched normal hepatic function participants to moderate hepatic impairment participants, received a single dose of firsocostat 20 mg (2 × 10 mg capsules) orally on Day 1.
- Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg: Matched normal hepatic function participants to severe hepatic impairment participants, received a single dose of firsocostat 5 mg (1 × 5 mg capsule) orally on Day 1.
- Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg: Matched normal hepatic function participants to mild hepatic impairment participants, received a single dose of fenofibrate 48 mg (1 × 48 mg tablet) orally on Day 1.
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
hr*ng/mL
  Firsocostat: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  Firsocostat | 160.6 (158.28) | 69.8 (38.73) | 682.1 (497.09) | 64.5 (33.22) | 310.4 (75.18) | 10.2 (2.92) |  |
  GS-834773: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  GS-834773 | 46.2 (57.67) | 7.4 (5.83) | 395.8 (535.93) | 5.1 (3.21) | 153.3 (65.72) | 1.4 (1.38) |  |
  Fenofibric Acid: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 10
  Fenofibric Acid |  |  |  |  |  |  | 61207.4 (24630.23) | 48128.0 (17377.69)
Statistical Analysis 1: Comparison: Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg vs Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg; AUClast of Firsocostat; Test type: Other; Geometric least-square mean (GLSM) ratio = 181, 90% CI 2-sided [98 to 332]
Statistical Analysis 2: Comparison: Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg vs Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg; AUClast of Firsocostat; Test type: Other; GLSM ratio = 881, 90% CI 2-sided [488 to 1589]
Statistical Analysis 3: Comparison: Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg vs Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg; AUClast of Firsocostat; Test type: Other; GLSM ratio = 3081, 90% CI 2-sided [2446 to 3881]
Statistical Analysis 4: Comparison: Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg vs Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg; AUClast of GS-834773; Test type: Other; GLSM ratio = 430, 90% CI 2-sided [185 to 998]
Statistical Analysis 5: Comparison: Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg vs Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg; AUClast of GS-834773; Test type: Other; GLSM ratio = 4417, 90% CI 2-sided [1867 to 10449]
Statistical Analysis 6: Comparison: Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg vs Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg; AUClast of GS-834773; Test type: Other; GLSM ratio = 14676, 90% CI 2-sided [7932 to 27153]
Statistical Analysis 7: Comparison: Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg vs Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg; AUClast of Fenofibric Acid; Test type: Other; GLSM ratio = 122, 90% CI 2-sided [86 to 173]

2. Primary Outcome: PK Parameter: AUCinf of Firsocostat, GS-834773 (Primary Metabolite of Firsocostat), and Fenofibric Acid (Primary Metabolite of Fenofibrate)
Description: AUCinf is defined as the concentration of drug extrapolated to infinite time. The PK of fenofibric acid was evaluated in participants with mild hepatic impairment and matched participants with normal hepatic function (Cohort 4).
Time Frame: as for outcome 1
Population: Participants in the PK Analysis Sets were analyzed. 6 participants with normal hepatic function served as matched controls across both Cohort 1 and 2.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
hr*ng/mL
  Firsocostat: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  Firsocostat | 165.2 (162.71) | 70.5 (38.82) | 686.6 (499.35) | 65.8 (34.36) | 313.6 (72.68) | 10.6 (2.97) |  |
  GS-834773: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  GS-834773 | 48.5 (59.21) | 8.2 (5.84) | 399.0 (537.09) | 5.9 (3.46) | 155.9 (65.85) | 1.6 (1.37) |  |
  Fenofibric Acid: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 10
  Fenofibric Acid |  |  |  |  |  |  | 65530.7 (25917.76) | 50754.1 (18262.73)
Statistical Analysis 1: Comparison: Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg vs Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg; AUCinf of Firsocostat; Test type: Other; GLSM ratio = 183, 90% CI 2-sided [100 to 337]
Statistical Analysis 2: Comparison: Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg vs Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg; AUCinf of Firsocostat; Test type: Other; GLSM ratio = 869, 90% CI 2-sided [482 to 1568]
Statistical Analysis 3: Comparison: Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg vs Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg; AUCinf of Firsocostat; Test type: Other; GLSM ratio = 2976, 90% CI 2-sided [2389 to 3708]
Statistical Analysis 4: Comparison: Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg vs Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg; AUCinf of GS-834773; Test type: Other; GLSM ratio = 399, 90% CI 2-sided [179 to 892]
Statistical Analysis 5: Comparison: Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg vs Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg; AUCinf of GS-834773; Test type: Other; GLSM ratio = 3843, 90% CI 2-sided [1641 to 9000]
Statistical Analysis 6: Comparison: Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg vs Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg; AUCinf of GS-834773; Test type: Other; GLSM ratio = 10712, 90% CI 2-sided [6525 to 17585]
Statistical Analysis 7: Comparison: Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg vs Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg; AUCinf of Fenofibric Acid; Test type: Other; GLSM ratio = 125, 90% CI 2-sided [89 to 174]

3. Primary Outcome: PK Parameter: Cmax of Firsocostat, GS-834773 (Primary Metabolite of Firsocostat), and Fenofibric Acid (Primary Metabolite of Fenofibrate)
Description: Cmax is defined as the maximum observed concentration of drug. The PK of fenofibric acid was evaluated in participants with mild hepatic impairment and matched participants with normal hepatic function (Cohort 4).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
ng/mL
  Firsocostat: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  Firsocostat | 50.9 (45.96) | 25.4 (20.44) | 197.7 (118.67) | 20.1 (12.09) | 73.8 (17.70) | 3.0 (1.56) |  |
  GS-834773: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  GS-834773 | 12.9 (16.08) | 2.3 (2.11) | 77.3 (56.03) | 1.4 (1.16) | 31.3 (14.66) | 0.5 (0.64) |  |
  Fenofibric Acid: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 10
  Fenofibric Acid |  |  |  |  |  |  | 2723.0 (1078.36) | 2451.0 (808.68)
Statistical Analysis 1: Comparison: Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg vs Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg; Cmax of Firsocostat; Test type: Other; GLSM ratio = 169, 90% CI 2-sided [87 to 326]
Statistical Analysis 2: Comparison: Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg vs Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg; Cmax of Firsocostat; Test type: Other; GLSM ratio = 905, 90% CI 2-sided [537 to 1526]
Statistical Analysis 3: Comparison: Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg vs Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg; Cmax of Firsocostat; Test type: Other; GLSM ratio = 2719, 90% CI 2-sided [1994 to 3708]
Statistical Analysis 4: Comparison: Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg vs Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg; Cmax of GS-834773; Test type: Other; GLSM ratio = 391, 90% CI 2-sided [163 to 942]
Statistical Analysis 5: Comparison: Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg vs Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg; Cmax of GS-834773; Test type: Other; GLSM ratio = 4470, 90% CI 2-sided [2170 to 9207]
Statistical Analysis 6: Comparison: Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg vs Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg; Cmax of GS-834773; Test type: Other; GLSM ratio = 9278, 90% CI 2-sided [4945 to 17407]
Statistical Analysis 7: Comparison: Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg vs Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg; Cmax of Fenofibric Acid; Test type: Other; GLSM ratio = 109, 90% CI 2-sided [81 to 146]

4. Primary Outcome: PK Parameter: % AUCexp of Firsocostat, GS-834773 (Primary Metabolite of Firsocostat), and Fenofibric Acid (Primary Metabolite of Fenofibrate)
Description: %AUCexp is defined as the percentage of AUC extrapolated between AUClast and AUCinf. The PK of fenofibric acid was evaluated in participants with mild hepatic impairment and matched participants with normal hepatic function (Cohort 4).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of AUC
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
percentage of AUC
  Firsocostat: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  Firsocostat | 2.54 (2.378) | 1.36 (1.222) | 0.63 (0.788) | 1.92 (1.645) | 1.35 (1.953) | 4.68 (2.671) |  |
  GS-834773: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  GS-834773 | 7.16 (7.997) | 13.16 (12.642) | 1.71 (1.889) | 13.59 (12.288) | 2.21 (2.288) | 25.94 (19.497) |  |
  Fenofibric Acid: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 10
  Fenofibric Acid |  |  |  |  |  |  | 7.11 (3.767) | 5.38 (2.758)

5. Primary Outcome: PK Parameter: Tmax of Firsocostat, GS-834773 (Primary Metabolite of Firsocostat), and Fenofibric Acid (Primary Metabolite of Fenofibrate)
Description: Tmax is defined as the time (observed time point) of Cmax. The PK of fenofibric acid was evaluated in participants with mild hepatic impairment and matched participants with normal hepatic function (Cohort 4).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
hours
  Firsocostat: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  Firsocostat | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 1.02] | 1.00 [1.00 to 2.00] | 1.50 [1.00 to 2.00] | 2.50 [1.00 to 3.00] |  |
  GS-834773: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  GS-834773 | 1.50 [1.00 to 2.00] | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 1.02] | 1.50 [1.00 to 2.00] | 2.00 [2.00 to 2.00] | 2.50 [1.00 to 3.00] |  |
  Fenofibric Acid: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 10
  Fenofibric Acid |  |  |  |  |  |  | 3.00 [3.00 to 4.00] | 2.50 [2.00 to 3.00]

6. Primary Outcome: PK Parameter: Clast of Firsocostat, GS-834773 (Primary Metabolite of Firsocostat), and Fenofibric Acid (Primary Metabolite of Fenofibrate)
Description: Clast is defined as the last observed quantifiable concentration of drug. The PK of fenofibric acid was evaluated in participants with mild hepatic impairment and matched participants with normal hepatic function (Cohort 4).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
ng/mL
  Firsocostat: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  Firsocostat | 0.20 (0.114) | 0.10 (0.042) | 0.26 (0.359) | 0.10 (0.047) | 0.23 (0.204) | 0.08 (0.017) |  |
  GS-834773: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  GS-834773 | 0.11 (0.051) | 0.12 (0.070) | 0.18 (0.104) | 0.11 (0.077) | 0.22 (0.185) | 0.07 (0.027) |  |
  Fenofibric Acid: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 10
  Fenofibric Acid |  |  |  |  |  |  | 133.04 (51.253) | 90.71 (33.405)

7. Primary Outcome: PK Parameter: Tlast of Firsocostat, GS-834773 (Primary Metabolite of Firsocostat), and Fenofibric Acid (Primary Metabolite of Fenofibrate)
Description: Tlast is defined as the time (observed time point) of Clast. The PK of fenofibric acid was evaluated in participants with mild hepatic impairment and matched participants with normal hepatic function (Cohort 4).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
hours
  Firsocostat: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  Firsocostat | 24.00 [24.00 to 72.00] | 24.00 [24.00 to 24.00] | 72.00 [48.00 to 96.00] | 24.00 [24.00 to 48.00] | 48.00 [47.97 to 72.00] | 16.00 [12.00 to 16.00] |  |
  GS-834773: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  GS-834773 | 24.00 [16.00 to 72.00] | 12.00 [10.00 to 16.00] | 48.02 [24.00 to 96.00] | 11.00 [10.00 to 16.00] | 36.04 [24.00 to 48.00] | 7.00 [6.00 to 8.00] |  |
  Fenofibric Acid: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 10
  Fenofibric Acid |  |  |  |  |  |  | 96.00 [72.00 to 96.17] | 84.25 [72.00 to 96.00]

8. Primary Outcome: PK Parameter: λz of Firsocostat, GS-834773 (Primary Metabolite of Firsocostat), and Fenofibric Acid (Primary Metabolite of Fenofibrate)
Description: λz is defined as the terminal elimination rate constant, estimated by linear regression of the terminal elimination phase of the log plasma concentration of drug versus time curve of the drug. The PK of fenofibric acid was evaluated in participants with mild hepatic impairment and matched participants with normal hepatic function (Cohort 4).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
1/hour
  Firsocostat: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  Firsocostat | 0.132 (0.1093) | 0.155 (0.0684) | 0.096 (0.0753) | 0.136 (0.0796) | 0.077 (0.0204) | 0.193 (0.0765) |  |
  GS-834773: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  GS-834773 | 0.133 (0.0948) | 0.214 (0.0942) | 0.105 (0.0916) | 0.209 (0.0918) | 0.103 (0.0543) | 0.300 (0.1379) |  |
  Fenofibric Acid: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 10
  Fenofibric Acid |  |  |  |  |  |  | 0.034 (0.0080) | 0.038 (0.0082)

9. Primary Outcome: PK Parameter: CL/F of Firsocostat, GS-834773 (Primary Metabolite of Firsocostat), and Fenofibric Acid (Primary Metabolite of Fenofibrate)
Description: CL/F is defined as the apparent oral clearance following administration of the drug. The PK of fenofibric acid was evaluated in participants with mild hepatic impairment and matched participants with normal hepatic function (Cohort 4).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/hour
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
mL/hour
  Firsocostat: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  Firsocostat | 259318.9 (239527.46) | 376896.2 (228676.47) | 59482.2 (63193.83) | 395572.3 (226508.90) | 16969.7 (5154.88) | 509793.4 (168681.93) |  |
  GS-834773: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  GS-834773 | 1467352.6 (1790413.18) | 3966285.6 (2982349.95) | 239748.5 (351882.41) | 4795605.6 (2952570.14) | 44379.6 (38793.78) | 4656562.3 (2689827.70) |  |
  Fenofibric Acid: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 10
  Fenofibric Acid |  |  |  |  |  |  | 909.4 (539.09) | 1060.8 (391.86)

10. Primary Outcome: PK Parameter: Vz/F of Firsocostat, GS-834773 (Primary Metabolite of Firsocostat), and Fenofibric Acid (Primary Metabolite of Fenofibrate)
Description: Vz/F is defined as the apparent volume of distribution of the drug. The PK of fenofibric acid was evaluated in participants with mild hepatic impairment and matched participants with normal hepatic function (Cohort 4).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
mL
  Firsocostat: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  Firsocostat | 2896998.5 (2176020.23) | 2846198.8 (2249997.50) | 592810.8 (318935.52) | 3797739.4 (2684509.46) | 230242.5 (92293.34) | 3079474.8 (1593778.35) |  |
  GS-834773: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  GS-834773 | 15576712.2 (19451521.66) | 19236747.1 (10816737.06) | 2126366.5 (2117217.85) | 23635388.6 (10179635.17) | 501512.3 (524040.62) | 20312673.6 (18230756.23) |  |
  Fenofibric Acid: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 10
  Fenofibric Acid |  |  |  |  |  |  | 25908.5 (9331.48) | 28290.3 (8476.01)

11. Primary Outcome: PK Parameter: t1/2 of Firsocostat, GS-834773 (Primary Metabolite of Firsocostat), and Fenofibric Acid (Primary Metabolite of Fenofibrate)
Description: t1/2 is defined as the estimate of the terminal elimination half-life of the drug. The PK of fenofibric acid was evaluated in participants with mild hepatic impairment and matched participants with normal hepatic function (Cohort 4).
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg: Participants with mild hepatic impairment received a single dose of firsocostat 20 mg (2 × 10 mg capsules) orally on Day 1.
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 1 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10 | 10
hours
  Firsocostat: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  Firsocostat | 5.23 [3.91 to 25.19] | 4.39 [3.73 to 6.78] | 11.20 [6.57 to 13.56] | 5.04 [4.00 to 11.02] | 9.54 [7.89 to 10.79] | 3.93 [2.55 to 4.93] |  |
  GS-834773: number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 0 | 0
  GS-834773 | 5.24 [3.44 to 25.28] | 3.32 [2.58 to 3.97] | 12.82 [4.13 to 17.25] | 3.28 [2.88 to 3.85] | 8.51 [6.84 to 9.19] | 2.49 [1.78 to 3.51] |  |
  Fenofibric Acid: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 10
  Fenofibric Acid |  |  |  |  |  |  | 21.33 [17.90 to 26.43] | 18.27 [15.73 to 21.34]

12. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (AEs)
Description: Treatment-emergent adverse events (TEAEs) were defined as 1 or both of the following:
  * Any AEs with an onset date on or after the study drug start date and no later than 30 days after permanent discontinuation of study drug. If the AE onset date is the same as the date of study drug start date then the AE onset time must be on or after the study drug start time. If the AE onset time is missing when the start dates are the same, the AE will be considered treatment emergent.
  * Any AEs leading to premature discontinuation of study drug.
Time Frame: First dose date plus 30 days
Population: Participants in the Safety Analysis Set were analyzed. 6 participants served as matched control across both Cohort 1 and 2.
Measure: Number; unit: percentage of participants
Groups:
- Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg: Matched normal hepatic function participants to severe hepatic impairment participants received a single dose of firsocostat 5 mg (1 × 5 mg capsule) orally on Day 1.
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 1 & 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg
Number analyzed (Participants) | 10 | 10 | 14 | 10 | 10 | 10 | 10
percentage of participants | 20.0 | 10.0 | 7.1 | 30.0 | 10.0 | 0 | 10.0

13. Secondary Outcome: Percentage of Participants Experiencing Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from predose at any postdose visit, up to and including the date of last dose of study drug plus 30 days for subjects who permanently discontinued study drug. The most severe graded abnormality from all tests was counted for each participant.
Time Frame: First dose date plus 30 days
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 1 & 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function): Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function): Fenofibrate 48 mg
Number analyzed (Participants) | 10 | 10 | 14 | 10 | 10 | 10 | 10
Percentage of participants | 100.0 | 90.0 | 50.0 | 100.0 | 50.0 | 90.0 | 60.0

ADVERSE EVENTS:
Time Frame: First dose date plus 30 days
Description: Participants in the Safety Analysis Set were analyzed. 6 participants served as matched control across both Cohort 1 and 2.
Arm/Group | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg | Cohort 1 & 2 (Normal Hepatic Function): Firsocostat 20 mg | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg | Cohort 3 (Normal Hepatic Function) Firsocostat 5 mg | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg | Cohort 4 (Normal Hepatic Function) Fenofibrate 48 mg
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/14 | 0/10 | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/14 | 0/10 | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 1/10 | 1/14 | 3/10 | 1/10 | 0/10 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (Mild Hepatic Impairment): Firsocostat 20 mg (N=10) | Cohort 2 (Moderate Hepatic Impairment): Firsocostat 20 mg (N=10) | Cohort 1 & 2 (Normal Hepatic Function): Firsocostat 20 mg (N=14) | Cohort 3 (Severe Hepatic Impairment): Firsocostat 5 mg (N=10) | Cohort 3 (Normal Hepatic Function) Firsocostat 5 mg (N=10) | Cohort 4 (Mild Hepatic Impairment): Fenofibrate 48 mg (N=10) | Cohort 4 (Normal Hepatic Function) Fenofibrate 48 mg (N=10)
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT02891408/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT02891408/SAP_001.pdf